CLINICAL TRIAL: NCT05099029
Title: A Phase III, Multiple-center, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy, Immunogenicity, and Safety of an Adjuvanted, Inactivated Enterovirus 71 (EV71) Vaccine in Healthy Infants and Children
Brief Title: A Study to Evaluate the Efficacy, Immunogenicity and Safety of an EV71 Vaccine in Healthy Infants and Children
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Enimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EV-BR1701
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Enterovirus Infections
Keywords: Foot-and-Mouth Disease; Vaccines; Hand, foot and mouth Disease; EV71 vaccine
MeSH Terms: conditions — Enterovirus Infections; Foot-and-Mouth Disease; Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV71 Vaccine (Experimental)
  Interventions: Biological: EV71 vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: EV71 vaccine — EV71 vaccine ([1 μg total protein + adjuvant 150 μg AI(OH)3] per dose) Two vaccinations at 28 days apart
  Arms: EV71 Vaccine
Biological: Placebo — Placebo ([ adjuvant 150 μg AI(OH)3] per dose) Two vaccinations at 28 days apart
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the EV71vaccine efficacy, immune response and safety profiles after two injections of the cell culture-based inactivated EV71 vaccine with adjuvant Al(OH)3 administrated in pediatric population aged 2 months to 6 years old.

DETAILED DESCRIPTION:
The clinical trial designed in this Study is a placebo-controlled, double-blinded Phase III and is aimed to evaluate the vaccine efficacy, safety, immunogenicity and immune persistence of cell culture-based inactivated EV71 vaccine in children age of 2 months to <6 years old. Two doses of Alum-adjuvanted 1.0 μg per dose of EV71 vaccine candidate will be administrated to subjects. The efficacy will be evaluated within a two year period after receiving 2-regimen vaccination by comparing the EV71-associated disease rates between the vaccine and placebo groups. Whereas, the immunogenicity will be assessed on Day 56 and Day 196, and the immune persistence will be evaluated on Day 392. Safety will be followed up to Day 392.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged from 2 months to 6 years old (i.e. >= 2 months old and < 7 years old) at the time of first vaccination.
2. Subject's guardians are able and willing to comply with study procedures and provide the signed informed consent.
3. Subject is able and can comply with the requirements of the protocol.
4. Subject with body temperature <= 38℃.

Exclusion Criteria:

1. Subject with previous known Enterovirus 71 (EV71) infection or investigational EV71 vaccination.
2. Subject with a history of herpangina, hand-foot-mouth disease, and acute hemorrhagic conjunctivitis associated with enterovirus infection in the past 30 days.
3. Subject with a history of hypersensitivity to vaccines, or a history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
4. Subject under 2 years old with gestation <34weeks or a birth weight <2200g.
5. History of epilepsy, seizures or non-febrile convulsions that may affect subject participation in the study in the opinion of the investigator.
6. Severe malnutrition or dysgenopathy at the screening visit.
7. Major congenital defects or serious chronic illness, including perinatal brain damage at the screening visit.
8. Subject diagnosed of having autoimmune disease (e.g., celiac disease, type I diabetes, lupus (SLE), juvenile dermatomyositis, scleroderma, juvenile idiopathic arthritis (JIA), immune (or idiopathic) thrombocytopenia purpura) that may affect subject participation in the study in the opinion of the investigator.
9. Bleeding disorder diagnosed by a doctor or significant bruising or hemostatic difficulties with IM injections or blood draws.
10. Any acute febrile illness 3 days prior to administrating the first vaccination.
11. Use of any investigational product (including drug, vaccine) within 30 days prior to vaccination or planned use during Visit 1 to Visit 4 (Day 0 to Day 196).
12. Administration of any vaccine within 14 days prior to each study vaccination.
13. Use of immunoglobulins or any blood products within 3 months prior to vaccination.
14. Chronic administration (defined as > 14 day of continuous use) of systemic immunosuppressants, other systemic immunomodulators, or systemic corticosteroids within 6 months prior to vaccination.
15. Any condition that in the opinion of the investigator may interfere with the evaluation of study objectives.
16. Subject with any confirmed or suspected immunodeficiency.

Ages: 2 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3982 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of Hand, Foot and Mouth disease caused by EV71 after the second vaccination. | From 28 days after the second vaccination to two year
  Evaluate the efficacy of EV71 vacccine against HFMD caused by EV71
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | 28 days after the second vaccination
  Evaluate the immunogenicity by the response rate

SECONDARY OUTCOMES:
The incidence rate of the severe complications and hospitalization of EV71 associated HFMD/HA disease after the second vaccination. | From 28 days after the second vaccination to two year
  1. Evaluate the efficacy of vaccination against the severe complications, including neurologic, pulmonary edema, and cardiorespiratory failure, of EV71 associated HFMD/HA diseases after completion of full vaccination.
  2. Evaluate the efficacy of vaccination against the hospitalization of EV71 associated HFMD/HA diseases after completion of full vaccination.
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 0,56,196,and 392
  1. Evaluate the immunogenicity of EV71 vaccine with two-dose regimen.
  2. Evaluate the immune persistence of EV71 vaccine with two-dose regimen.
  3. Evaluate lot-to-lot consistency by comparing the immunogenicity induced by 3 independent EV71 vaccines.
Adverse events of EV71 vaccine | Day 0 to Day 392
  1. Occurrence and severity of solicited injection site relations and general reactions within 7 days following each injection.
  2. Occurrence and severity of unsolicited adverse events within 28 days following each injection.
  3. Occurrence and relations with vaccination of some special AE during the 6-months follow-up period (up to Day 196).
  4. Occurrence and relations with vaccination of serious adverse events (SAEs) during the one year follow-up period (up to Day 392).

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Fen Yang, Study Director — Enimmune Corporation
Locations (8):
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital HsinChu Branch, Hsinchu
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Pasteur Institute of HCMC, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided